CLINICAL TRIAL: NCT02279810
Title: Knowledge, Attitude and Practice About Organ Transplantation Among Medical Students and Medical Staff
Brief Title: Attitudes About Organ Transplantation
Acronym: KAPsurvey
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: International Institute of Rescue Research and Education (Other)
Responsible Party: Principal Investigator, Lukasz Szarpak, Lukasz Szarpak, International Institute of Rescue Research and Education
Other Study IDs: KAPtransplant2014
Record Dates: First submitted 2014-10-26; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Transplantation, Organ
Keywords: organ shortage; attitudes to organ transplantation
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Medical students, medical staff: Survey about Knowledge, Attitude and Practice About Organ Transplantation
  Interventions: Behavioral: survey

INTERVENTIONS:
Behavioral: survey — Survey

SUMMARY:
The study evaluates the knowledge, attitude and practice about organ transplantation among medical students and medical staff.

DETAILED DESCRIPTION:
Globally, almost every second a transplanted kidney comes from a living donor (LDTx); in Europe it is 18.1%, but in Poland it is only 2% (0.6 for 1 million from living donors). The number of patients awaiting on kidney transplantation (KTx) is increasing, and the number of deceased donors is constantly at a low level. This disturbing situation should motivate the entire interdisciplinary health team to seek new solutions.

In the study the investigators are examining how medical students and medical staff feel about the issues of organ transplantation, especially: organ shortage, cost of organ transplantation, definition of brain death.

The investigators are planning to focus on the following specific questions:

What is the level of knowledge about organ donation among participants? What are the sociodemographic, sociocultural and socioeconomic characteristics of listed as an Organ Donor and non-listed as an Organ Donor among medical staff and medical students? Evidence on the role of financial and other incentives in eliciting organ donation.

ELIGIBILITY:
Inclusion Criteria:

* Give voluntary consent to participate in the study

Exclusion Criteria:

* Not meet the above criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical staff: medical doctors, nurses, paramedics Medical students: PhD students, medicine students, nursing and paramedics studies
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2014-10; Primary Completion 2014-11 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who approve prosocial motivation to organ donation | 2 months
  Percentage of healthcare workers and medical students with appropriate attitude assessed by 10- items questionnaire about perception towards financial and other incentives in eliciting organ donation. For each correct answer participant receive 1 point (0-1 point scale).

SECONDARY OUTCOMES:
Results of the Medical Knowledge Tool (Questionnaire) | 2 months
  Percentage of healthcare workers and medical students with appropriate knowledge assessed by 10- items questionnaire about basic information about organ registry and qualification to transplantation. For each correct answer participant receive 1 point (0-1 point scale).
Results of the Practice Tool (Questionnaire) | 2 months
  Percentage of healthcare workers and medical students with appropriate practice assessed by 10- items questionnaire about basic information about practice with organ donation (prohibited and unethical practices). For each correct answer participant receive 1 point (0-1 point scale).

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Principal Investigator — National Institute of Cardiology, Warsaw, Poland; Lukasz Czyżewski, Principal Investigator — Medical University of Warsaw; Andrzej Kurowski, Principal Investigator — National Institute of Cardiology, Warsaw, Poland
Locations (2):
- Poland (2):
  - International Institute of Rescue Research and Education, Warsaw, Masovia
  - International Institute of Rescue Research and Education, Warsaw

REFERENCES:
- [Background] Czyzewski L, Wyzgal J. The adequacy of transplantation education in the ESRD population in Poland. Ann Transplant. 2012 Apr-Jun;17(2):62-73. doi: 10.12659/aot.883224. PMID 22743724